CLINICAL TRIAL: NCT00331110
Title: Immediate and Short-Term Analgesic and Biomechanical Effects of a Laterally Wedged Insole With Ankle Strapping for Medial Compartment Knee Osteoarthritis
Brief Title: Study of How An Ankle Strap Changes Effects of Insole Treatment for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Physiatric Association of Spine, Sports and Occupational Rehabilitation (Other); Foundation for Physical Medicine and Rehabilitation (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200501707
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2007-04

CONDITIONS: Medial Compartment Knee Osteoarthritis

INTERVENTIONS:
Device: Laterally-Wedged Insole with Ankle Strapping
Device: Laterally-Weged Insole

SUMMARY:
The goal of this project is to assess the effects of an ankle strap on the effectiveness of a laterally-wedged insole with ankle strapping in reducing knee symptoms and improving static and dynamic lower limb biomechanics. Using a repeated measures, modified cross-over design, the following aims and hypotheses will be addressed:

Biomechanical Hypotheses

1. Use of the insole with ankle strapping significantly alters hip-knee-ankle (HKA) angle towards 180° or talar valgus angulation.
2. Use of the insole with ankle strapping significantly reduces peak knee external varus moment during gait.
3. Use of the insole with ankle strapping significantly reduces foot external rotation (out-toeing) or widened base during gait analysis.
4. The radiographic HKA angle and tilt angle of the talus will predict knee peak external varus moment during gait.

Clinical Hypotheses

1. The use of an insole with ankle strapping over a two-week period will reduce knee pain (Visual analogue scale, and Knee Osteoarthritis Outcome Survey).

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is a common cause of pain and disability and the medial compartment is involved most frequently. If conservative mechanical therapies could reduce knee OA symptoms, risks to patients might be minimized through reduction in use of pharmacotherapy or surgery. A lateral heel wedge with strapping of the ankle joint has been reported to induce a similar therapeutic effect to that of proximal tibial osteotomy. It is presumed that the mechanism for this involves correction of genu varum. However, the effects on the static lower limb mechanical axis and the dynamic knee adduction moment, a risk factor for knee OA symptoms and progression, have not been assessed, so the mechanism of effect is currently unknown. The proposed protocol would compare lower limb mechanical alignment (measured by radiographic hip-knee-ankle angle) and dynamic knee varus moment (measured by 3-dimensional gait analysis) with and without the strapped insole to further understanding of the mechanism of effect on subjects with knee OA. Additionally, this protocol would assess analgesia and whether use of the insole reduces known knee joint unloading compensatory mechanisms during gait. Through measurement of radiographic lower limb alignment, dynamic knee varus moment, and ankle/foot static and dynamic angles, a model would be developed relating radiographs with dynamic moments, potentially allowing greater risk stratification for knee OA development and progression through use of radiographs. In addition to elucidating the mechanism of effect of this insole and developing a model for radiographic interpretation, this protocol would be the fist study of this insole involving non-Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 45 or over will be included if they have predominantly medial compartment knee OA by American College of Rheumatology criteria, with medial knee pain rated at least 40/100mm on a visual analogue scale on most days of the month during one of the past 3 months.

Exclusion Criteria:

* Potential subjects with a body mass index (BMI) of greater than 35 will be excluded to avoid the potential confounding effect of increased weight on the height of the insole. Other exclusion criteria will include: known injury or surgery involving bone or cartilage of the knee or ankle which may alter gait, history of factors which might alter response to use of a laterally wedged insole (e.g. greater or similar reduction in lateral compared with medial femorotibial jont space width on posterior-anterior radiographs, tibial osteotomy, congenital foot problems, fused joints, foot deformity, known limitation of range of motion of the subtalar joint), known neuromuscular disease, co-morbid disease which might confound gait analysis (e.g. hip OA, ankle OA, hallux rigidus, valgus deformity of the midfoot, other symptomatic deformity of the foot, advanced arthroplasty of the hindfoot, previous ankle arthrodesis, unable to walk without a gait aid), current use of an orthotic insole, inability to comply with study protocol.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 2006-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Hip-Knee-Ankle Alignment
Talar Tilt Angle
External Knee Adduction Moment
Pain Assessment
Gait Velocity

SECONDARY OUTCOMES:
Center of Pressure
Foot Progression Angle

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States